CLINICAL TRIAL: NCT04964583
Title: Double-blind, Randomized, Prospective, Parallel Study to Demonstrate the Efficacy and Safety of Outpatient Treatment of the Fixed Combination of Hydroxychloroquine With Azithromycin Versus Hydroxychloroquine Treatment and Placebo Treatment in Patients Diagnosed With Mild COVID-19 Infection
Brief Title: Hidroxicloroquina With Azitromicina Versus Hidroxicloroquina and Placebo Int Patients With Mild COVID-19
Acronym: Omehecatl
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Ultra Laboratorios SA. de CV. (Unknown)
Responsible Party: Principal Investigator, Rodolfo Rivas Ruiz, MD, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-785-138
Record Dates: First submitted 2021-06-25; First posted 2021-07-16 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydroxychloroquine with Azithromycin (Experimental): Fixed combination of Hydroxychloroquine with Azithromycin 200 mg / 250 mg one tablet every 12 hours for five days and continue with Hydroxychloroquine 200 mg one tablet every 12 hours for 5 more days.
  Interventions: Drug: Hydroxychloroquine with Azithromycin
- Hydroxychloroquine (Active Comparator): Hydroxychloroquine 200 mg, one tablet every 12 hours for ten days.
  Interventions: Drug: Hydroxychloroquine with Azithromycin
- Placebo (Placebo Comparator): Placebo one tablet every 12 hours for ten days.
  Interventions: Drug: Hydroxychloroquine with Azithromycin

INTERVENTIONS:
Drug: Hydroxychloroquine with Azithromycin — Fixed combination of Hydroxychloroquine with Azithromycin 200 mg / 250 mg one tablet every 12 hours for five days and continue with Hydroxychloroquine 200 mg one tablet every 12 hours for 5 more days.
  Other Names: Azithromycin

SUMMARY:
Chloroquine and hydroxychloroquine are two antimalarial drugs that are also used in autoimmune diseases. Chloroquine analogs have been shown to inhibit endosome acidification and exhibit nonspecific antiviral activity at high micromolar concentration in vitro against a wide range of emerging viruses (HIV, dengue, hepatitis C, chikungunya, influenza, Ebola, SARS, and MERS ). virus) and more recently COVID-19. On the other hand, azithromycin is a macrolide antibiotic indicated for infections caused by sensitive pathogens, but which in combination with Hydroxychloroquine has shown a synergistic effect against the SARS-CoV-2 virus.

International studies show the lack of beneficial effect in hospitalized or mechanically ventilated patients. Referring that because these medications reduce the in case of having a beneficial effect it would be in the early onset, to avoid inflammation (cytokine storm), and thus prevent hospitalizations.

The present study focuses on characterizing the possible synergy of the fixed combination of hydroxychloroquine associated with azithromycin in the treatment of Covid-19 from mild to moderate manifestations. Three treatment schemes are proposed with a 10-day follow-up, a) the fixed combination of Hydroxychloroquine / Azithromycin (combination of interest), b) Hydroxychloroquine (active comparison group) and c) non-active control group, using placebo. A group of patients between 18 and 75 years old is considered, who may or may not present other comorbidities. Follow-up will be carried out through quantification of viral load, evaluation of the systemic inflammatory state, changes in clinical manifestations and possible effect on the reduction of hospitalizations. Therefore, it is proposed to carry out the following project.

objective To determine the efficacy and safety of Hydroxychloroquine / Azithromycin fixed combination compared to Hydroxychloroquine or placebo in outpatients with Research design: Phase II, multicenter, prospective, randomized, parallel, longitudinal, double-blind study.

Medications to use Group 1. Fixed combination of Hydroxychloroquine with Azithromycin 200 mg / 250 mg one tablet every 12 hours for five days and continue with Hydroxychloroquine 200 mg one tablet every 12 hours for 5 more days.

Group 2. Hydroxychloroquine 200 mg, one tablet every 12 hours for ten days. Group 3. Placebo one tablet every 12 hours for ten days.

ELIGIBILITY:
Inclusion Criteria:

* Have given the signed informed consent form.
* Confirmed diagnosis of COVID-19 infection by PCR with mild symptoms.
* Patients who attend the primary care respiratory care module in the participating units and who have symptoms suggestive of COVID-19, who comply with the current operational definition.
* With or without comorbidities such as hypertension, controlled diabetes mellitus, cardiovascular or respiratory diseases.
* Controlled diabetes will be considered to be that which is evidenced by results of glycosylated hemoglobin less than 7% in the last 3 tables, whether it is reported in your beneficiary file or by external laboratory results.
* Electrocardiogram (ECG) normal or with variations without clinical relevance, with QT interval <450 ms.
* No contraindication to study drugs (history of hypersensitivity to study drugs, including macrolides, patients with renal failure (eGFR <40 mL / min) or on renal replacement therapy, patients with a history of retinopathy or macular degeneration.

Exclusion Criteria:

* Patients who are participating in studies with investigational drugs.
* Pregnancy or breastfeeding.
* Type 1 diabetes
* % Type II diabetes mellitus with glycated hemoglobin greater than 7%.
* Patients requiring hospitalization or assisted mechanical ventilation
* Cardiac disorders with cardiac conduction delay (QT segment ≥ 450 ms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Hospitalization | 15 days
  Being admitted for hospitalization

SECONDARY OUTCOMES:
Viral load | 0 and 14 days
  Measured by RT-PCR
Clinical safety | 21 days
  any adverse event

CONTACTS AND LOCATIONS:
Locations (3):
- Mexico (3):
  - UMF 28, Benito Juárez, Mexico City
  - Fundación IMSS, Cuauhtémoc, Mexico City
  - UMF 52, Cuautitlán Izcalli, State of Mexico

IPD SHARING:
Plan to Share IPD: Yes
Database with all non identifiable data will be available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months